CLINICAL TRIAL: NCT05494411
Title: Named Patient Program for Mitomycin for Pyelocalyceal Solution
Status: Available | Type: Expanded Access
Sponsor: UroGen Pharma Ltd. (Industry)
Collaborators: Tanner Pharma Group (Other)
Responsible Party: Sponsor
Other Study IDs: UT003
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Urothelial Cancer of Renal Pelvis; Urothelial Carcinoma of the Renal Pelvis and Ureter; Urothelial Carcinoma Ureter; Urothelial Carcinoma Ureter Recurrent; Urothelial Carcinoma; Urothelial Carcinoma Recurrent
Keywords: Low-grade Upper Tract Urothelial Cancer; LG-UTUC; UGN-101; Mitomycin
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Mitomycin

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Mitomycin for pyelocalyceal solution
  Other Names: JELMYTO

SUMMARY:
This program provides controlled, pre-approval access to JELMYTO in response to unsolicited requests by physicians, hospitals, pharmacies, distributors, ministries of health or other parties on behalf of specific, or named patients, in select countries where JELMYTO has not yet received a marketing authorization and in situations when patients have exhausted all available treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are suitable to receive JELMYTO and for whom there is reasonable expectation that JELMYTO may provide clinical benefit based on the medical judgment of their prescribing physician.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult